CLINICAL TRIAL: NCT02751671
Title: Are Stimulated Clean-Catch Urine Collection Techniques More Successful When Combined With Prior Emergency Point-of-care Ultrasound in Paediatric Patients?
Brief Title: Point-of-care Ultrasound for Clean-Catch Urine Collection in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Jocelyn Gravel, MD, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: POCUS CCU
Record Dates: First submitted 2016-04-21; First posted 2016-04-26 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-04

CONDITIONS: Urinalysis; Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- POCUS before clean catch sampling (Experimental): The intervention of interest will be the use of emergency point-of-care ultrasound performed by a research assistant to evaluate bladder fullness before clean-catch stimulation manoeuvre. More specifically, following randomisation, children in the experimental group will have ePOCUS to measure the transversal bladder diameter. If the transversal bladder diameter is > 2 cm, the CCU procedure will be started without a prior feeding period. If the diameter is < 2 cm, the CCU will be postponed for a 20 minute feeding period and a new ePOCUS will be done. After the second ePOCUS, the CCU will be done if the transversal bladder diameter reaches > 2cm. If not, the child will have another 20 minute feeding period and a third ePOCUS prior to proceeding to the CCU regardless the bladder diameter.
  Interventions: Procedure: POCUS
- Standard clean catch sampling (Experimental): Patients allocated to this arm will have a 20 minute feeding period either being breastfed or provided with formula intake appropriate to the infant's age and weight. If possible, the genital areas of the infant will be cleaned with warm water and soap and dried with sterile gauze prior to the feeding. The parents will let the diaper opened and will be will be ready to collect urine if the child voids during the feeding period. After the feeding, the stimulated clean-catch procedure will be performed without prior ultrasound
  Interventions: Procedure: Standard

INTERVENTIONS:
Procedure: POCUS — The use of Point-of-care ultrasound before urine sample procedure
  Arms: POCUS before clean catch sampling
Procedure: Standard — Urine sampling procedure without prior ultrasound
  Arms: Standard clean catch sampling

SUMMARY:
Background:

The investigators recently evaluated a new bladder stimulation technique to obtain clean-catch urine in infants aged less than six months. In this study, the reported success rate was of 52%. Measuring the transversal bladder diameter prior to the procedure with emergency point-of-care ultrasound (ePOCUS) could likely increase success rates for this technique as it has been described for bladder scans prior to performing urethral catheterization.

Objective:

The aim of this study is to evaluate if using emergency point-of-care ultrasound to measure bladder volume improves clean-catch urine collection success in patients less than 6 months of age when compared to children undergoing this technique without a prior ultrasound.

Methods:

This will be a randomized controlled trial performed in a tertiary paediatric emergency department. Participants will include all infants younger than 6 months of age who need a urinary culture and/or analysis requested by the attending physician. The intervention will consist of the use of emergency point-of-care ultrasound by a trained research assistant. The primary outcome will be the rate of success of the procedure. Secondary objectives will be to evaluate time to collect urine samples and to determine which transversal bladder diameter correlates with more than a 90% success rate for the procedure. Independent variables will be sex and age. In both groups, trained research nurses will collect clean-catch urine samples using bladder stimulation techniques. The success rate of the CCU procedure in both groups will be calculated. The time required to collect urine samples will be analysed. In group 1, the investigators will determine the transversal bladder diameter corresponding to a success rate for the procedure of > 80%. It is estimated that, in the worse-case scenario, the evaluation of 200 participants will provide a 95% confidence interval smaller than 10% for proportions. In addition, 20 participants with a successful CCU sample would allow to evaluate 2 risk factors using univariate and multivariate analysis.

Expected results:

This study will demonstrate that use of emergency point-of-care ultrasound increases success rates of stimulated clean-catch manoeuvres and may avoid invasive urethral catheterizations in young children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged less than 6 months
* Urine sample ordered by the treating physician
* Presence of a research assistant

Exclusion Criteria:

* Any medical condition where obtaining a midstream urine sample is impossible (e.g. urostomy, anuria for 24h)
* Any serious illness or unstable infant (e.g. sepsis)
* Any medical situation where the infant cannot be fed (e.g NPO order, GCS<15)
* Inability to obtain parental informed consent (language barrier, absence, etc.)

Max Age: 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 201 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Successful clean-catch manoeuver | 5 minutes
  The rate of successful clean-catch urine sample collection. Success is defined by the collection of a sample of urine of at least 2 mL, obtained within 300 seconds of bladder stimulation manoeuvers or obtained while disinfecting prior to the manoeuvre.

SECONDARY OUTCOMES:
Delay for collection | 1 hour
  Time to collect urine sample from randomisation to sample collection
delay for procedure | 1 hour
  Time to collect urine sample from beginning of stimulation to sample collection
Nurse time | 2 hours
  Time that nurses have to spend with the patients

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weill O, Labrosse M, Levy A, Desjardins MP, Trottier ED, Gravel J. Point-of-care ultrasound before attempting clean-catch urine collection in infants: a randomized controlled trial. CJEM. 2019 Sep;21(5):646-652. doi: 10.1017/cem.2019.30. PMID 31006399